CLINICAL TRIAL: NCT00806923
Title: A Randomized, Double-blind Study of the Effect of Avastin Plus Cisplatin and Gemcitabine or Placebo Plus Cisplatin and Gemcitabine on Progression-free Survival in Treatment-naïve Patients With Advanced or Recurrent Non-squamous NSCLC
Brief Title: A Study of Avastin (Bevacizumab) in Patients With Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO17704
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Cisplatin; Gemcitabine; Bevacizumab

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: bevacizumab [Avastin]
- 2 (Experimental)
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: bevacizumab [Avastin]
- 3 (Placebo Comparator)
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Placebo

INTERVENTIONS:
Drug: Cisplatin — 80mg/m2 iv on day 1 of each 3 week cycle, for a maximum of 6 cycles
Drug: Gemcitabine — 1250mg/m2 on days 1 and 8 of each 3 week cycle for a maximum of 6 cycles
Drug: Placebo — iv on day 1 of each 3 week cycle until disease progression
  Arms: 3
Drug: bevacizumab [Avastin] — 15mg/kg 1v on day 1 of each 3 week cycle until disease progression
  Arms: 1
Drug: bevacizumab [Avastin] — 7.5 mg/kg iv on day 1 of each 3 week cycle until disease progression
  Arms: 2

SUMMARY:
This 3 arm study will evaluate the efficacy and safety of adding Avastin versus placebo to a standard chemotherapeutic regimen in patients with advanced or recurrent non-squamous non-small cell lung cancer (NSCLC) who have not received prior chemotherapy. The anticipated time of study treatment is until disease progression, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* documented inoperable, locally advanced, metastatic or recurrent non-squamous NSCLC;
* adequate liver and kidney function;
* women of childbearing potential must have a negative serum pregnancy test within 7 days of starting study treatment.

Exclusion Criteria:

* prior chemotherapy or treatment with another systemic cancer therapy;
* surgery (including open biopsy), significant traumatic injury, or radiotherapy within the last 4 weeks prior to first dose of study treatment;
* brain metastasis or spinal cord compression;
* fertile men, and women of childbearing potential, not using adequate contraception;
* treatment with any other investigational agent, or participation in another clinical trial, within 30 days prior to entering the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1044 (Actual)
Dates: Start 2005-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Event driven

SECONDARY OUTCOMES:
Efficacy: Duration of overall survival, time to treatment failure, response rate, and duration of response. | Event driven
Safety:AEs, laboratory tests, SAEs, coagulation parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (122):
- Argentina (5):
  - Bahía Blanca
  - Buenos Aires
  - Mendoza
  - San Miguel de Tucumán
  - Santa Fe
- Australia (10):
  - Adelaide
  - Brisbane
  - Canberra
  - Kurralta Park
  - Melbourne
  - Parkville
  - Perth
  - Sydney
  - Tugun
  - Wollongong
- Belgium (4):
  - Brussels
  - Haine-Saint-Paul
  - Leuven
  - Liège
- Brazil (4):
  - Belo Horizonte
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- Bulgaria (5):
  - Plovdiv
  - Sofia
  - Stara Zagora
  - Varna
  - Veliko Tarnovo
- Canada (11):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Victoria, British Columbia
  - Moncton, New Brunswick
  - London, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Sainte-Foy, Quebec
- Czechia (3):
  - Ostrava
  - Prague
  - Ústí nad Labem
- France (13):
  - Belfort
  - Bobigny
  - Caen
  - Lyon
  - Marseille
  - Montbéliard
  - Montpellier
  - Pierre-Bénite
  - Rennes
  - Rouen
  - Saint-Herblain
  - Strasbourg
  - Vandœuvre-lès-Nancy
- Germany (12):
  - Berlin
  - Essen
  - Gauting
  - Göttingen
  - Hamburg
  - Heidelberg
  - Hemer
  - Karlsruhe
  - Leverkusen
  - Mainz
  - Mannheim
  - München
- Greece (3):
  - Alexandroupoli
  - Athens
  - Thessaloniki
- Hong Kong, Hong Kong
- Hungary (6):
  - Budapest
  - Mosdós
  - Nyíregyháza
  - Székesfehérvár
  - Szombathely
  - Zalaegerszeg
- Israel (5):
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Italy (10):
  - Candiolo
  - Catania
  - Genova
  - Milan
  - Napoli
  - Parma
  - Perugia
  - Reggio Emilia
  - Roma
  - Rozzano
- Poland (7):
  - Gdansk
  - Gdynia
  - Lublin
  - Olsztyn
  - Poznan
  - Szczecin
  - Warsaw
- Russia (3):
  - Balashikha
  - Moscow
  - Saint Petersburg
- Spain (9):
  - Alicante
  - Barakaldo
  - Barcelona
  - Girona
  - Madrid
  - Málaga
  - San Cristóbal de La Laguna
  - Seville
  - Valencia
- Taiwan (3):
  - Kueishan
  - Taichung
  - Taipei
- Thailand (2):
  - Bangkok
  - Chiang Mai
- United Kingdom (6):
  - Guildford
  - London
  - Manchester
  - Sheffield
  - Sutton
  - Yeovil

REFERENCES:
- [Derived] Leighl NB, Bennouna J, Yi J, Moore N, Hambleton J, Hurwitz H. Bleeding events in bevacizumab-treated cancer patients who received full-dose anticoagulation and remained on study. Br J Cancer. 2011 Feb 1;104(3):413-8. doi: 10.1038/sj.bjc.6606074. Epub 2011 Jan 18. PMID 21245868
- [Derived] Leighl NB, Zatloukal P, Mezger J, Ramlau R, Moore N, Reck M, Manegold C. Efficacy and safety of bevacizumab-based therapy in elderly patients with advanced or recurrent nonsquamous non-small cell lung cancer in the phase III BO17704 study (AVAiL). J Thorac Oncol. 2010 Dec;5(12):1970-6. doi: 10.1097/JTO.0b013e3181f49c22. PMID 20978447
- [Derived] Reck M, von Pawel J, Zatloukal P, Ramlau R, Gorbounova V, Hirsh V, Leighl N, Mezger J, Archer V, Moore N, Manegold C; BO17704 Study Group. Overall survival with cisplatin-gemcitabine and bevacizumab or placebo as first-line therapy for nonsquamous non-small-cell lung cancer: results from a randomised phase III trial (AVAiL). Ann Oncol. 2010 Sep;21(9):1804-1809. doi: 10.1093/annonc/mdq020. Epub 2010 Feb 11. PMID 20150572